CLINICAL TRIAL: NCT01280448
Title: The Correlation Between Lung Cancer Susceptibility, Drug Response and Genetic Polymorphism
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Department of Hematology-oncology, WanFang Hospital
Other Study IDs: 99054
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Tobacco Smoking; gene polymorphism
MeSH Terms: conditions — Lung Neoplasms; Tobacco Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — genes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case Group
- Control Group

SUMMARY:
Lung cancer is the leading cause of cancer deaths in Taiwan. The carcinogen in the environment is a key role in the development of lung cancer, and one of its main resource is tobacco. Activated carcinogens in the organism lead to mutations of crucial oncogenes resulting in tumor development. Genes such as Cytochrome P-450 family, GST (glutathione S-transferase) family, UGT (UDP-Glucuronosyltransferase) family, ERCC-1(excision repair cross-complementing rodent repair deficiency),ERCC-4 and ERCC-5,are encoding antioxidant enzymes or involving in the DNA repair process and the production of some transcription factors. In recent years, many studies have shown the correlation between these genes and the susceptibility of lung cancer. Each gene has a different role in the tumor development pathway. CYP, UGT, GST, NAT2 (N-acetyltransferase 2) and NQO1(NAD(P)H:quinono oxidoreductase 1) involve in the production of antioxidant enzymes. The antioxidant enzymes can detoxificate hydrogen peroxide or defense against oxidative stress. However, the genetic polymorphisms may influence the function of detoxification, which cause the increase in the susceptibility of lung cancer. P53 and MDM2 genes play important roles in the production of tumor-suppression proteins and the regulation of transcription factors, which may regulate the growth and the apoptosis of cell cycle and influence the susceptibility of lug cancer. The polymorphisms in ERCC genes may cause the damage in the DNA repair process which might also cause increase in lung cancer susceptibility. The overexpression of epidermal growth factor receptor is highly correlated with increasing risk of the non-small cell lung cancers. The overexpression may induce the proliferation of cancer cells and the inhibition of the apatosis. Therefore, in recent years, EGFR has been widely studied as the new target of the drugs and the susceptibility of the lung cancer. In addition,the genetic polymorphisms in drug metabolism channel proteins, like OCT2 (organic cation transporter), ATP7A, ATP7B and ABC (ATP-binding cassette) transporter may have influence on the metabolism, the efficacy and the toxicity of the drugs.

DETAILED DESCRIPTION:
The current study is a matched case-control study. The experimental group is the patients diagnosed as lung cancer at Taipei Medical University- Wanfang Hospital from January 2010 to December 2013, and one healthy patient will be matched to each case as the control group. The purpose of the current study is to investigate the association between genetic polymorphisms and lung cancer in the Taiwanese population and to analyze the correlation.

ELIGIBILITY:
Inclusion Criteria:

* This study has two groups, the case group and the control group. The match criteria is patients with the same gender and the age is ± 5 years.

  1. Case group - Patients with the pathology diagnosed as the primary lung cancer patients.
  2. Control group - Patients without any cancer or disease history of cancers.

Exclusion Criteria:

* Case group - Patients with the pathology diagnosed as the non-primary lung cancer patients or the patients with lung cancer induced by other cancer metastasis.
* Control group -

  1. With other cancers.
  2. With COPD induced by smoking or the genetic factors.
  3. With familial adenomatous polyposis
  4. With HIV infection, hepatitis B or hepatitis C

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2010-09; Study Completion 2013-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Gjin Eugene Liu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan